CLINICAL TRIAL: NCT04798131
Title: Treat Refractory Auditory Hallucinations in Schizophrenia Patients With fMRI-guided Neurofeedback: a Randomized-controlled Trial
Brief Title: fMRI-based Neurofeedback to Relieve Drug-resistant Auditory Hallucinations
Acronym: INTRUDE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: National Research Agency, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020_08; 2020-A00631-38 (Other: ID-RCB number,ANSM); ANR-16-CE37-0015 (Other: ANR number)
Record Dates: First submitted 2021-01-14; First posted 2021-03-15 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Schizophrenia; Hallucinations, Auditory; Hallucinations, Visual
Keywords: Schizophrenia; Hallucinations; Drug-resistance; functional MRI; Neurofeedback; Machine-Learning.
MeSH Terms: conditions — Schizophrenia; Hallucinations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): The visual feedback will correspond to instructions, adapted to the current hallucinatory state and decoded online from the fMRI signal.
  Interventions: Other: Active neurofeedback procedure
- Sham (Sham Comparator): The visual feedback will correspond to random instructions independently of the fMRI signal.
  Interventions: Other: Sham neurofeedback procedure

INTERVENTIONS:
Other: Active neurofeedback procedure — Patients will perform 5 fMRI sessions. Four consecutive fMRI runs (1/ day) during which they will continuously receive visual feedback computed from the fMRI signal analyzed with the hallucinations decoder. Patients will be trained to maintain the brain state associated with the no-hallucination state using appropriate coping strategies. A 5th fMRI scan will be performed at 1 month post-treatment.
  Arms: Active
Other: Sham neurofeedback procedure — Patients will perform 5 fMRI sessions. Four consecutive fMRI runs (1/ day) during which they will receive a random feedback and a 5th run at 1 month post-treatment.
  Arms: Sham

SUMMARY:
The INTRUDE trial aims at assessing the efficacy of an fMRI-based neurofeedback procedure on drug-resistant auditory hallucinations. Hallucinations are complex and transient mental states associated with subtle and brain-wide patterns of activity for which we were recently able to validate an fMRI multivariate decoder. Based on this progress, we can track patients' hallucinatory status using real-time fMRI. We will test whether schizophrenia patients with drug-resistant hallucinations can be trained to maintain the brain state associated with a no-hallucination condition using appropriate strategies and thus reduce overall severity. We will refer to a double-blind randomized placebo-controlled design. A total of 86 patients will be enrolled and equally split in an active neurofeedback group (n=43) and a sham group (n=43), matched for sex, age and PANSS scores. Each patient will benefit from 4 runs of either active or sham neurofeedback. The primary outcome measure will be the mean decrease of AHRS scores relative to baseline, and at 1 month post-treatment. We expect significant clinical benefits from fMRI-based neurofeedback on drug-resistant hallucinations compared with the sham group.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia (according to the DSM-5 classification)
* Frequent auditory hallucinations (SAPS item #1 ≥ 4)
* Stable medication for at least 30 days
* Absence of chronic neurological disorder (including seizure)
* Able to provide free written consent to participate in the research

Exclusion Criteria:

* Pregnancy
* Contraindication to MRI scan
* Claustrophobia
* No social insurance

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Auditory Hallucination Rating Scale (AHRS) measure of hallucinations severity | 1 month after treatment
  AHRS will be measured at t0 (randomization) and at 1 month after treatment Minimum score is 2, maximum score is 41, higher score indicates more severe symptoms.

SECONDARY OUTCOMES:
Change from baseline in Positive and Negative Syndrome Scale (PANSS) measure of hallucinations severity | 1 month after treatment
  PANSS will be measured at t0 (randomization) and at 1 month after treatment The PANSS contains 7 positive symptom scales, 7 negative system scales, and 16 general psychopathology symptom scales. rate from 1 to 7 on each symptom scale. The total score is the sum of all scales with a minimum score of 30 and a maximum score of 210
Change from baseline Questionnaire for Psychotic Experiences (QPE) measure for severity of hallucinations | 1 month after treatment
  QPE will be measured at t0 (randomization) and at 1 month after treatment
Change from baseline Simplified Acute Physiology Score (SAPS) measure for severity of hallucinations | 1 month after treatment
  SAPS will be measured at t0 (randomization) and at 1 month after treatment
Change from baseline Visual analogue scale (VAS) measure for severity of hallucinations | 1 month after treatment
  VAS will be measured at t0 (randomization) and at 1 month after treatment
Changes in global functioning relative to baseline | 1 month after treatment
  Global Assessment of Functioning (GAF) is a numeric scale be measured at t0 (randomization) and at 1 month after treatment Scores range from 100 (extremely high functioning) to 1 (severely impaired).
Changes in quality of life relative to baseline | 1 month after treatment
  SQLS score will be measured at t0 (randomization) and at 1 month after treatment
Changes in structural MRI markers relative to baseline | 1 month after treatment
  Cortical thickness will be measured at t0 (randomization) and at 1 month after treatment
Changes in structural MRI markers relative to baseline | 1 month after treatment
  Gyrification Index will be measured at t0 (randomization) and at 1 month after treatment
Changes in functional MRI markers relative to baseline | 1 month after treatment
  Brain activity at rest and connectivity metrics will be measured at t0 (randomization) and at 1 month after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Renaud JARDRI, MD,PhD, Principal Investigator — University Hospital, Lille